CLINICAL TRIAL: NCT02084524
Title: ANC1 Study Impact of a Geriatric and Nutritional Evaluation for the Malnutrition and Malnutrition Risk Screening in Patients Over 70 Years With Colorectal Surgery.
Acronym: ANC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2011.703
Record Dates: First submitted 2013-11-04; First posted 2014-03-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Tumor
Keywords: vulnerable; nutrition; cancer; colorectal; tumor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutritional evaluation (No Intervention)
  Interventions: Procedure: Malnutrition screening and perioperative nutritional support

INTERVENTIONS:
Procedure: Malnutrition screening and perioperative nutritional support — * Multidisciplinary training sessions for malnutrition and malnutrition risk screening, postoperative nutritional procedures according to the ESPEN Guidelines
  * Preoperative Geriatric evaluation : eligibility criteria, nutritional status, previous history, comorbidities, clinical examination, activities of daily living (ADL) and Instrumental activities of daily living (IADL)
  * Implementation of an adapted nutritional support based on ESPEN Guidelines

SUMMARY:
Malnutrition priori a major abdominal surgery is frequent and increases morbidity and mortality. The management of malnutrition has an impact in reducing postoperative complications. However malnutrition is rarely detected and Guidelines infrequently followed.

Recovery time and nutritional evaluation in elderly patients are major criteria in their postoperative management. Identifying malnutrition or malnutrition risk is fundamental to its treatment. It is therefore unsurprising that many validated tools for nutrition risk screening and nutrition assessment exist for the clinician to use in assisting with the accurate identification, referral and treatment of patients who are malnourished or at risk of malnutrition.

And nutritional management must be adapted and based on this evaluation and evolution of the general status (Guidelines Grade A).

A geriatric evaluation based on a screening of preoperative malnutrition should allow a better implementation of the European Society of Parenteral and Enteral Nutrition (ESPEN) guidelines.

DETAILED DESCRIPTION:
Assessing the impact of a geriatric action (Team Mobile Geriatrics, EMG, or if the geriatric facility team when it does not have EMG) on the rate of nutritional support perioperative elderly subjects (≥ 70 years) who underwent a colorectal cancer according to ESPEN recommendations and SFNEP.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 70 years
* Colorectal or tumor resection with/without synchronous metastases

Exclusion Criteria:

* Emergency resection of colorectal tumor
* Unresectable colorectal tumor with/without synchronous metastases

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative nutritional management | During perioperative period From D-7 before date of hospitalization until discharge from the hospital, up to 30 days
  Rate of nutritional support implemented in accordance with current European guidelines (ESPEN)

SECONDARY OUTCOMES:
Malnutrition screening | During preoperative seven days
  Rate of malnutrition screening procedure
Rate of preoperative nutritional management by immunonutrition implemented | During preoperative seven days
  Nutritional management by immunonutrition implemented is based on a complete nutritional evaluation
Rate of malnourished patients | During preoperative seven days
  Rate of malnourished patients is defined by the ESPEN criteria
Rate of patients with cachexia | Seventh day preoperative
  Rate of patients with cachexia is defined by the French National Authority for Health (HAS) criteria
Postoperative complications | Postoperative follow-up until discharge from hospital, up to 30 days
  Rate and type of postoperative complications (Grade I, II et IIIa of Dindo classification)
Rate of postoperative nutritional management implemented | Postoperative follow-up until discharge from hospital, up to 30 days
  Nutritional management implemented is based on the ESPEN guidelines
Evolution of the activities of daily living | During preoperative seven days and postoperative follow-up until discharge from hospital, up to 30 days
  Variations of Activities of daily living (ADL) and Instrumental activities of daily living (IADL) scores

CONTACTS AND LOCATIONS:
Locations (1):
- Professeur Marc BONNEFOY, Pierre-Bénite, France

REFERENCES:
- [Derived] Dupuis M, Kuczewski E, Villeneuve L, Bin-Dorel S, Haine M, Falandry C, Gilbert T, Passot G, Glehen O, Bonnefoy M. Age Nutrition Chirugie (ANC) study: impact of a geriatric intervention on the screening and management of undernutrition in elderly patients operated on for colon cancer, a stepped wedge controlled trial. BMC Geriatr. 2017 Jan 7;17(1):10. doi: 10.1186/s12877-016-0402-3. PMID 28061830